CLINICAL TRIAL: NCT02811146
Title: Cardiac Rehabilitation and Noninvasive Ventilation in Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, BRUNA THAYS SANTANA DE ARAÚJO, physiotherapist, clinical research, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 54735716.3.0000.5208
Record Dates: First submitted 2016-06-02; First posted 2016-06-23 (Estimated); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Heart Failure
Keywords: Heart Failure; Noninvasive Ventilation; Positive- Pressure Respiration
MeSH Terms: conditions — Heart Failure | interventions — Continuous Positive Airway Pressure; Cardiac Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Cardiopulmonary exercise testing (Experimental): Assess whether people who wore noninvasive ventilation during aerobic exercise have greater functional capacity than those who did not wear.
  Interventions: Device: Bilevel Positive Pressure Airway; Other: Heart rehabilitation
- ADL Glitre test (Experimental): Check that people who wore noninvasive ventilation during aerobic exercise have greater submaximal functional capacity than those who did not wear. Compare a ventilatory metabolic response of the ADL Glitre test with an six-minute walk test. .
  Interventions: Device: Bilevel Positive Pressure Airway; Other: Heart rehabilitation
- Minnesota Living with Heart Failure (Experimental): Check if people undergoing heart rehabilitation has improved quality of life.
  Interventions: Device: Bilevel Positive Pressure Airway; Other: Heart rehabilitation
- Bioimpedance balance (Experimental): Check if people undergoing heart rehabilitation has improved the body composition.
  Interventions: Device: Bilevel Positive Pressure Airway; Other: Heart rehabilitation
- Six-minute walk test (No Intervention): Compare a ventilatory metabolic response of the six-minute walk test with an ADL Glitre test.
- Metabolic ventilatory response (Experimental): To verify if non-invasive ventilation during aerobic exercise modifies the ventilatory metabolic response in patients with heart failure.
  Check the metabolic ventilatory response during the Glittre ADL test and six-minute walk test.
  Interventions: Device: Bilevel Positive Pressure Airway; Other: Heart rehabilitation

INTERVENTIONS:
Device: Bilevel Positive Pressure Airway — Heart rehabilitation with noninvasive ventilation, for 12 weeks, 3 times a week
  Arms: ADL Glitre test; Bioimpedance balance; Cardiopulmonary exercise testing; Metabolic ventilatory response; Minnesota Living with Heart Failure
Other: Heart rehabilitation — Heart rehabilitation, for 12 weeks, 3 times a week
  Arms: ADL Glitre test; Bioimpedance balance; Cardiopulmonary exercise testing; Metabolic ventilatory response; Minnesota Living with Heart Failure

SUMMARY:
The study aims to demonstrate the efficacy of NIV continuously in cardiac rehabilitation programs, improvement of exercise tolerance, with consequent reflection in functional capacity and quality of life of this population.

DETAILED DESCRIPTION:
BACKGROUND: Heart failure (HF) is a cardiovascular syndrome with enormous impact on public health by high morbidity and mortality rates that are associated. Studies show that changes in striated skeletal muscle of those individuals, possibly caused by progressive physical inactivity, contribute to the construction of the pathophysiology of this disease, emphasizing the importance of exercise for these patients. Exercise programs can be traced safer and related form the actual functional capacity thereof. Cardiac rehabilitation it is a set of activities that aims to ensure that patients with heart disease the best conditions, especially physical. In this context, non-invasive ventilation (NIV) is an alternative to provide an improved tolerance during exercise in patients with HF.

GOALS: Evaluate the effectiveness of the use of NIV association to aerobic exercise in exercise programs supervised during cardiac rehabilitation exercise tolerance and quality of life in patients with heart failure when compared to performing these exercises without ventilatory support.

METHODS: This is a clinical trial, controlled, randomized and blind to be developed with patients arising out of the main Recife reference centers in the care of patients with heart failure. It will be conducted assessments of functional capacity made by cardiopulmonary exercise testing (CPET), the Glittre-ADL test and through the questionnaire Duke Activity Status Index (DASI), assessment of quality of life using the questionnaire Minnesota Living with Heart Failure (MLWHF), and finally, in order to determine a clinical change, will be used to Patient Global Impression of Change Scale (PGIS).

EXPECTED RESULTS: This study aims to demonstrate the efficacy of NIV continuously in cardiac rehabilitation programs, improvement of exercise tolerance, with consequent reflection in functional capacity and quality of life of this population.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary adults diagnosed with heart failure of ischemic hypertensive or alcoholic etiology;
* Ejection fraction of the left ventricle smaller than 50% (LVEF <50%) assessed by echocardiography simple;
* Recent and functional class II and III by the New York Heart Association (NYHA);
* FEV1 <80% predicted and / or FEV1 / FVC> 70% predicted;
* Clinical stability; Ex-smokers for more than five years;
* No change in the class of drugs within three months prior to the beginning of the study.

Exclusion Criteria:

* Patients with unstable angina;
* Myocardial infarction or heart surgery up to three months before the survey;
* FEV1 / FVC <70% predicted characterizing obstructive respiratory disorder;
* Respiratory diseases;
* Smoking;
* Hemodynamic instability;
* Trauma of recent face;
* Nausea and vomiting;
* Orthopedic and neurological diseases;
* Psychic changes that restrict them to respond to the questionnaire.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07; Primary Completion 2021-05-31 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary exercise testing | Baseline and 12 weeks
  Change in functional capacity
Glittre-ADL Test | Baseline and 12 weeks
  Change in submaximal functional capacity
Six-Minute Walk Test | Baseline
  Change in submaximal functional capacity
Ventilatory metabolic response during the 6-minute walk test (6MWT) and Glittre-ADL Test | Baseline and 12 weeks
  Compare the ventilatory metabolic response of the six-minute walk test and Glittre-ADL Test

SECONDARY OUTCOMES:
Minnesota Living with Heart Failure | Baseline and 12 weeks
  Improved in quality of life
Bioimpedance scale | Baseline and 12 weeks
  Change in the body composition

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Hospital of the Clinics Federal University of Pernambuco, Recife, Pernambuco
  - Cardiopulmonary Physiotherapy Laboratory, Recife, Pernambuco

IPD SHARING:
Plan to Share IPD: Undecided